CLINICAL TRIAL: NCT02564835
Title: Effects of Yoga on Cognitive and Immune Function in Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Oncology Nursing Society (Other)
Responsible Party: Principal Investigator, Moira Visovatti, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00096913
Record Dates: First submitted 2015-09-23; First posted 2015-10-01 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Yoga; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research assistants at Time 2 and 3 are blinded to which arm the participant is in.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Yoga (Experimental): The Yoga Program includes two 90-minute classes every week tor a total of 12 weeks.
  Interventions: Other: Yoga
- Physical Activity (Active Comparator): The Physical Activity Program includes two 90-minutes classes every week for a total of 12 weeks.The intervention is based on the Exercise for People Living with Cancer program and will include nine resistance exercises (e.g. standing push up, squats, standing leg curl) and 8 flexibility exercises (e.g. shoulder stretch, quadriceps stretch, hamstrings and lower back stretch) targeted for the whole body as well as a brief warm up and cool down (walking).
  Interventions: Other: Physical Activity
- Usual Care (No Intervention): Participants randomized to this arm will receive standard care only.

INTERVENTIONS:
Other: Yoga — The yoga curriculum in this study is based is based on the Integral Yoga approach that includes branches of yoga associated with cognitive and immune benefits (Hatha, Raja). Within the Integral Yoga approach, physical poses, breathing techniques and mediation practices were chosen to provide benefits to the nervous system, immune system, musculoskeletal system and gastrointestinal system. Poses will be adapted to individual needs. The number of repetitions and/or length of hold will be increased through standard progression.
  Arms: Yoga
Other: Physical Activity — The physical activity intervention is based on the Exercise for People Living with Cancer program. The intervention will include nine resistance exercises (e.g. squats) and 8 flexibility exercises (e.g. shoulder stretch) targeted for the whole body as well as a brief warm up and cool down (walking). Exercises will be adapted to individual needs. The number of repetitions and/or length of hold will increase through standard progression.
  Arms: Physical Activity

SUMMARY:
The purpose of this study is to determine if individuals with colorectal cancer enjoy yoga and to begin to assess whether yoga is effective in improving attention and immune function in individuals with colorectal cancer compared to physical activity and usual care.

DETAILED DESCRIPTION:
The proposed study will use a prospective RCT pilot design with three arms (yoga, resistance and flexibility exercise, usual care) and a total of 60 men and women who have completed therapy (> 6 months post primary or adjuvant therapy) to accomplish the specific aims. Equal numbers of men and women will be randomized into each arm of the study. Participants will be tested before, immediately after, and 3-months after treatment or similar time points for the usual care group. After data has been collected, participants who were randomized to the resistance and flexibility exercise group (active control group) or to the usual care group will be provided with the opportunity to participate in the yoga intervention.

ELIGIBILITY:
Inclusion Criteria:

* a history of any stage new or recuurent colorectal cancer
* great then 6 months post treatment for colorectal cancer
* report not fully recovered from the effects of cancer and cancer treatment
* no clinical signs or symptoms of brain metastasis
* normal (or corrected to normal) hearing and vision
* able to read and write English

Exclusion Criteria:

- conditions that could affect participation in yoga such as spinal disease or unstable joints

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Program Evaluation | At the end of the 12-week yoga and physical activity programs.
  The program evaluation was developed by the investigator to measure the participant experience and satisfaction with the interventions.

SECONDARY OUTCOMES:
Attention Network Test | Change from baseline to 6 months.
  The Attention Network Test is a computerized test that asks participants to determine the direction of an arrow in the center of the screen (left or right). The center arrow can be located above or below the center fixation and is accompanied by flankers and cues. Overall attention and the three networks are assessed by measuring accuracy and response times for correct answers and how response times for correct answers are influenced by flankers, alerting cues, and spatial cues.
Digit Span | Change from baseline to 6 months
  Digit Span asks participants to repeat a series of numbers in the order they were given (Digit Span Forward) or reverse order (Digit Span Backward). The score is the number of digits recalled in the correct order before two failed trials. Digit Span is a test of attention and cognitive control.
Digit Symbol Substitution Test | Change from baseline to 6 months
  The Digit Symbol Substitution Test provides participants with a key of numbers associated with symbols and ask participants to fill in numbered blank squares with the appropriate symbol. The score is the number of blank square filled in within 120 seconds. Digit Symbol Substitution test is a test of attention and cognitive control.
Trail Making Test | Change from baseline to 6 months
  The Trail Making Test asks participants to draw a line connecting numbered circles (Part A) and a line connecting numbered circles and letters (Part B). The score is the time taken to complete the task. The Trail Making Test is a test of attention and cognitive control.
Attentional Function Index | Change from baseline to 6 months
  The Attentional Function Index is a questionnaire that asks participants to rate their function on everyday tasks requiring attention and cognitive control from 0 (not at all) to 10 (extremely well or a great deal). The score is the average of 13 questions. The internal consistency ranges from 0.76 to 0.94 in individuals with cancer.
Functional Assessment of Cancer Therapy - Cognitive Function | Change from baseline to 6 months
  The Functional Assessment of Cancer Therapy-Cognitive Function is a questionnaire that measures perceived cognitive function and impact on quality of life from 0 (not at all) to 4 (very much). It includes 27 items grouped into 5 subscales The internal consistency is 0.96 on each subscale in individuals with cancer.
Pro-inflammatory Markers | Change from baseline to 6 months
  Serum levels of interleukin-1 beta, tumor necrosis factor-alpha, interleukin-6, interleukin-8, interleukin-12, interleukin-1 receptor antagonist, soluble tumor necrosis factor-receptor II, and c-reactive protein will be determined by cytometric bead array assay on a Luminex analyzer (MPXHYCTO-60K, Millipore; LXSAH, R & D Systems). Serum levels of neopterin will be determined by enzyme-linked immunosorbent assay (RE59821, IBL International). Blood samples will be collected between 8 am and 10 am.

OTHER OUTCOMES:
Attendance Log | Throughout the 12-week program.
  The attendance log was developed by the investigator to measure adherence to the intervention and dose of the intervention received. Participants sign the attendance log at each yoga or physical activity class
Adherence and Attrition Log | From date of signed informed consent until last yoga/physical activity class or research visit - up to 6 months
  The adherence and attrition log was developed by the investigator to describe reasons for not attending a class or dropping out of study. Participants will be asked if they would like to tell research team reason for missing a class or dropping out (e.g. too busy) so we can improve the intervention.
Safety Log | At each yoga and physical activity class throughout the 12-week program
  The safety log was developed by the investigator to describe any adverse event related to the yoga and physical activity programs.
Demographic and Medical Information Questionnaires | At baseline before randomization to study arm
  The demographic and medical information questionnaires were developed by the investigator to describe sample characteristics (such as age and stage of disease).
Profile of Mood States-Brief Form | Change from baseline to 6 months
  The Profile of Mood States-Brief Form asks participants to rate how they have been feeling (e.g. tense) in the past week on a scale of 0 (not at all) to 4 (extremely). The anxiety and depressed mood subscales will be used to describe the sample. Each subscale has five items and the score is the sum of the five items. The internal consistency of the anxiety and depressed mood subscales range from 0.86 to 0.93 in individuals with cancer.
Mindful Attention Awareness Scale | Changes from baseline to 6 monts
  The Mindful Attention Awareness Scale will be used to assess cognitive training or uptake of the yoga intervention. The questionnaire has 15 items and measures the frequency of mindful states in cancer.
Beliefs about Treatment | Changes from baseline to end of 12-week intervention
  The Benefits about Treatment Question was developed by investigators at University of California, Los Angeles to assess a participant's expectations about the yoga and physical activity interventions and their effect on outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Moira Visovatti, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Nursing, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No